CLINICAL TRIAL: NCT05256277
Title: A Phase 1 Study of Evaluating Preliminary Safety and Efficacy of CT101a in the Treatment of Relapsed or Refractory (r/r) AML Patients
Brief Title: NK Cell Therapy for AML
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: A new study is planed to replace the current study due to IP upgrade
Sponsor: Zhejiang University (Other)
Collaborators: Shanghai Zeke Biotechnology Co.，Ltd (Unknown)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT101a-001
Record Dates: First submitted 2022-02-08; First posted 2022-02-25 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: AML
Keywords: cytokine-induced memory-like NK cells; relapsed or refractory acute myeloid leukemia
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT101a (Experimental): 1 dose infusion
  Interventions: Drug: CT101a

INTERVENTIONS:
Drug: CT101a — cytokine-induced memory-like NK cells

SUMMARY:
This is a single-arm, open-label, non-randomized, multiple-dose, phase 1 dose escalation study evaluating the safety, efficacy and PK of CT101a in patients with relapsed/refractory acute myeloid leukemia.

Primary Objective:

To evaluate the safety and tolerability of CT101a and estimate the MTD in Chinese patients.

Secondary Objective:

To determine the preliminary efficacy of CT101a in the treatment of r/r AML by IWG response rate; To determine the duration of response, time to progression, disease-free survival, and overall survival of AML patients treated with CT101a.

Exploratory Objective:

To investigate and analyze the correlation between the donor KIR gene and the efficacy in the subject.

To explore the feasibility and safety of multiple doses of CT101a in the treatment of r/r AML.

To detect blood samples and bone marrow samples before and after CT101a infusion by single cell sequencing method, and to perform difference analysis.

DETAILED DESCRIPTION:
This is a single-arm, open-label, non-randomized, multiple-dose, phase 1 dose escalation study evaluating the safety, efficacy and PK of CT101a in patients with relapsed/refractory AML.

This clinical study is to evaluate the safety, MTD and preliminary efficacy of CT101a in patients with relapsed/refractory AML. Up to 9-18 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with relapsed or refractory AML:

   1. For patients with relapsed AML: after complete response (CR), leukemia cells or blast cells in the bone marrow reappear >5% (except for other reasons such as bone marrow regeneration after consolidation chemotherapy).
   2. For patients with refractory AML: initial cases who have been treated with standard regimens for 2 courses of treatment that are not effective; after CR, they undergo consolidation and intensive treatment and relapse within 12 months; those who relapse after 12 months but are ineffective after conventional chemotherapy; those who relapse for 2 or multiple times.
   3. AML patients with disease progression after transplantation.
2. Male or female ≥ 18 years old.
3. ECOG Performance Status 0 to 2.
4. Life expectancy ≥3 months.
5. Available HLA-haploidentical donor meeting the following criteria:

   1. Related donor (parent, sibling, offspring, or offspring of sibling);
   2. At least 18 years of age;
   3. HLA-haploidentical donor/recipient match by at least Class I serologic typing at the A&B locus;
   4. In general, the donor is healthy and can tolerate leukapheresis for collecting NK cells required in this study;
   5. Negative for HCV antibody, five items of HBV, HIV antibody and syphilis on donor viral screening;
   6. The female donor of childbearing potential must have a negative pregnancy test within screening.
   7. Voluntary written consent to participate in this study.
6. Adequate organ function as defined below:

   1. Total bilirubin<2 mg/dL;
   2. AST(SGOT)/ALT(SGPT) <3.0 x ULN;
   3. Creatinine within normal institutional limits;
   4. Oxygen saturation ≥90% on room air;
   5. Ejection fraction ≥35%.
7. Able to be off corticosteroids and any other immune suppressive medications beginning on 3 days before the CT101a infusion and continuing until 28 days after the CT101a infusion. However, use of low-level corticosteroids is permitted at the judgment of the investigator if deemed medically necessary. Low-level corticosteroid use is defined as 10mg or less of prednisone (or equivalent for other steroids) per day.
8. Women of childbearing potential must have a negative pregnancy test within screening. Female and male patients (along with their female partners) must agree to use two forms of acceptable contraception, including one barrier method, during participation in the study.
9. Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

1. Acute or chronic GVHD with ongoing active systemic treatment.
2. Circulating blast count >30,000/μL by morphology or flow cytometry.
3. Prior treatment with ML NK cell therapy within 3 months prior to screening.
4. Patients who are undergoing any approved or investigational chemotherapy and anti-leukemic therapy with small molecule-targeted drugs within the 14 days prior to the first dose of fludarabine.
5. Presence of any severe or uncontrolled systemic disease or condition.
6. Patients with active infection requiring systemic therapy within 2 weeks prior to screening.
7. HBsAg positive and HBV DNA is detectable or above the cut-off value or positive HCV antibody or positive HIV antibody or positive syphilis test.
8. New progressive pulmonary infiltrates on screening chest X-ray or chest CT scan that have not been evaluated with bronchoscopy.
9. Patients with a significant cardiovascular disease or condition.
10. Inadequate bone marrow reserve or organ function.
11. Other patients judged inappropriate for this study by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
DLT/MTD | 28 days
  The severity of adverse events is graded according to NCI-CTCAE version 5.0, and the investigator will determine whether the subject has DLT.
  Taking into account the clinical characteristics of AML patients, DLT is defined as: During the 28-day DLT observation period after CT101a infusion, the subject still has any of the following conditions related to the study drug despite the treatment measures taken:
  1. Non-hematology related DLT: Any non-hematologic AE ≥ Grade 3 that is caused by CT101a treatment and does not resolve to below Grade 2 within 3 days; infusion-related reactions will not be considered as DLT.
  Patients with clinical progression of AML after CT101a infusion can receive cytoreductive therapy (such as hydroxyurea, cytarabine) to control their disease, and maintain the DLT assessment during the entire DLT period, but any AE related to cytoreductive therapy will not be considered as DLT.

SECONDARY OUTCOMES:
Safety parameters | 2 years
  adverse events (AEs), serious adverse events (SAEs), laboratory test abnormalities, ECG changes and vital signs, physical examination abnormalities, etc.
overall response rate | 2 years
  The overall response rate (ORR, CR+CRi+PR) after cell infusion
DOR | 2 years
  DOR is defined as the time from the first date of the tumor achieving CR or CRi, until the first date of disease progression or death from any cause
OS | 2 years
  OS is defined as the time from the date of CT101a infusion until death from any cause
TTP | 2 years
  TTP is defined as the time from the date of CT101a infusion until the first date of leukemia progression.
LFS | 2 years
  LFS is defined as the time from the date of CT101a infusion until the first date of leukemia progression or relapse or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Huang He, PhD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affiliated Hospital，College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China